CLINICAL TRIAL: NCT03175471
Title: Cross-sectional Study for Assessment of MRI Based Biomarkers of Bile Duct Injury and Hepatic Fibrosis in Pediatric Onset Autoimmune Liver Disease
Brief Title: MRI Based Biomarkers in Pediatric Autoimmune Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN001-MRI biomarkers in AILD
Record Dates: First submitted 2017-01-31; First posted 2017-06-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Liver Disease; Primary Sclerosing Cholangitis; Autoimmune Hepatitis
MeSH Terms: conditions — Cholangitis, Sclerosing; Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum samples, Liver biopsy tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with autoimmune liver disease: Patients (6-23 y.o.) with established clinical diagnosis of AIH or suspected diagnosis of AIH based on elevated serum AST or ALT, elevated IgG level >1.1 ULN, elevated titer of autoantibodies, including ANA, SMA, LKM, LC-1 or SLA, which is consistent with the simplified criteria for the diagnosis of AIH in children will be enrolled.
  Patients (6-23 y.o.) with established clinical diagnosis of PSC or Suspected diagnosis of PSC supported by abnormal cholangiogram (ERCP or MRCP) or elevated GGT>1.5 ULN and dilated bile ducts by liver ultrasound will be enrolled.

SUMMARY:
Autoimmune liver diseases (AILD), which include Primary Sclerosing Cholangitis (PSC) and Autoimmune Hepatitis (AIH) are a common etiological factors for chronic liver disease among adolescents. In all these conditions, autoimmune lymphocyte responses are thought to orchestrate inflammatory injury against hepatocytes (primarily in AIH) or cholangiocytes (in PSC). In this proposal we aim to evaluate the Magnetic Resonance Imaging (MRI) modalities; MR cholangiopancreatography (MRCP) and MR elastography (MREL), as non-invasive biomarkers to assess two primary pathophysiological processes of AILD: bile duct damage and liver fibrosis. In this cross-sectional study MRI based findings of bile duct injury and liver fibrosis will be correlated with both liver histology and circulating biomarkers of these disease processes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-23 years old.
2. Established or suspected clinical diagnosis of AIH or PSC.

Exclusion Criteria:

1. History of liver transplantation.
2. Chronic Hepatitis B or untreated hepatitis C virus infection.
3. Pregnancy.
4. Absolute contraindication for MRI (e.g. pacemaker, metallic implants, claustrophobia).
5. Diagnosis of cystic fibrosis or biliary atresia
6. Diagnosis of cardiac hepatopathy.
7. Diagnosis of Wilson's disease, Alpha-1 Antitrypsin deficiency, or Glycogen storage disease.
8. Skin conditions which could be aggravated by MREL (i.e. Epidermolysis bullosa).

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 115 patients between 6 and 23 years of age with a diagnosis of PSC or AIH will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
MRI based outcomes | 36 months
  MRCP based assessment of intrahepatic and extrahepatic duct irregularities by Majoie classification (on 4 and 5 point scale of 0-3 and 0-4 respectively; 0: No visible abnormalities, 1: minimal dilatation/irregularities, 2: saccular dilatations/segmental stricture, 3: severe pruning, 4: Extremely irregular margin).
  MREL based quantification of mean shear stiffness (kPa) of liver.
Liver histopathology based assessment of bile duct injury by ISHAK Score | 36 months
  Assessment of bile duct injury by ISHAK Score (Confluent necrosis: on the 7 point scale of 0-6; Focal necrosis on the 4 point scale of 0-4 and portal inflammation on the 4 point scale of 0-4).
Liver histopathology based assessment of bile duct injury by Ludwig score | 36 months
  Assessment of bile duct injury by Ludwig score (on five point scale of 0-4; 0: No ductal injury, 1: portal inflammation, 2: periportal inflammation, 3: Portal bridging, 4: Nodular cirrhosis).
Liver histopathology based assessment of liver fibrosis by Nakanuma score | 36 months
  Assessment of liver fibrosis by Nakanuma score for on the 4 point scale of 0-3 (0; No portal fibrosis, 1; Portal fibrosis; 2; Bridging fibrosis, 3; Liver cirrhosis) .
Liver histopathology based assessment of liver fibrosis by Ishak score | 36 months
  Assessment of liver fibrosis by Ishak score on the 7 point scale of 0-6 (0; Absent, 1; confluent necrosis, 2; necrosis in some areas, 3; necrosis in most areas, 4; necrosis with occasional portal-central bridging necrosis, 5; necrosis with multiple portal-central bridging necrosis, 6; Panacinar or multiacinar necrosis).
Liver histopathology based assessment of cholangitis and hepatic activity | 36 months
  Cholangitis and hepatic activity by Nakanuma score for on the 4 point scale of 0-3 (0; No bile duct loss, 1; Bile duct loss in <1/3 of portal tracts; 2; Bile duct loss in 1/3-2/3 of portal tracts, 3; Bile duct loss in >2/3 of portal tracts).
Serum based outcome | 36 months
  Quantification of serum alkaline phosphatase (ALP in U/L) and Gamma-glutamyl transpeptidase (GGT in U/L).
Enhanced Liver Fibrosis (ELF) score | 36 months
  Assesment of Enhanced Liver Fibrosis (ELF) score on continuous scale of 1-10; <7.7 none -mild. ≥7.7 -<9.8 moderate, >9.8 sever).

SECONDARY OUTCOMES:
MR T1rho, T1, T2 Imaging | 36 Months
  Mean of MR T1rho, T1, T2 signal in msec to measure the inflammation.
Liver Morphometry | 36 Months
  Collagen deposition in percent area fibrosis by image analysis
Liver histopathology based outcomes | 36 Months
  Liver histopathology based grade of inflammation by Scheuer score on 5 point scale of 0-4; (0: No ductal injury, 1: portal inflammation, 2: periportal inflammation, 3: Portal to portal bridging, 4: Nodular cirrhosis).
Serum based outcomes | 36 Months
  Quantification of serum fractionated ALP (U/L)
Serum MMP7 | 36 Months
  Quantification of serum MMP7 (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Miethke, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahalingam N, Trout AT, Zhang B, Castro-Rojas C, Miethke AG, Dillman JR. Longitudinal changes in quantitative magnetic resonance imaging metrics in children and young adults with autoimmune liver disease. Abdom Radiol (NY). 2023 Jun;48(6):1933-1944. doi: 10.1007/s00261-022-03733-9. Epub 2023 Feb 17. PMID 36799997
- [Result] McCrary J, Trout AT, Mahalingam N, Singh R, Rojas CC, Miethke AG, Dillman JR. Associations Between Quantitative MRI Metrics and Clinical Risk Scores in Children and Young Adults With Autoimmune Liver Disease. AJR Am J Roentgenol. 2022 Jul;219(1):142-150. doi: 10.2214/AJR.21.27204. Epub 2022 Jan 26. PMID 35080454
- [Result] Dillman JR, Trout AT, Taylor AE, Khendek L, Kasten JL, Sheridan RM, Sharma D, Karns RA, Castro-Rojas C, Zhang B, Miethke AG. Association Between MR Elastography Liver Stiffness and Histologic Liver Fibrosis in Children and Young Adults With Autoimmune Liver Disease. AJR Am J Roentgenol. 2024 Jul;223(1):e2431108. doi: 10.2214/AJR.24.31108. Epub 2024 Apr 17. PMID 38630086